CLINICAL TRIAL: NCT04193215
Title: A Study of V114 and Acute Otitis Media in Children (PNEU-ERA)
Brief Title: V114 and Acute Otitis Media (V114-032/PNEU-ERA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-032; V114-032 (Other: MSD); 2023-001146-11 (EudraCT Number)
Record Dates: First submitted 2019-12-09; First posted 2019-12-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Otitis Media (AOM)
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive an intramuscular (IM) injection.
  Interventions: Biological: V114; Other: Pediatric vaccines
- Control (Other)
  Interventions: Other: Pediatric vaccines

INTERVENTIONS:
Biological: V114 — IM injection
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Other: Pediatric vaccines — Standard of care vaccines administered according to the local recommended schedule.

SUMMARY:
The primary objective is to evaluate V114 in the prevention of vaccine-type acute otitis media (VT-AOM) and the safety of V114 with respect to the proportion of participants with serious adverse events (SAEs) through completion of the study. The primary hypothesis is that V114 is superior to no V114 in preventing VT-AOM as assessed by the incidence of VT-AOM.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy (based on a review of medical history and physical examination)
* Is male or female, approximately 2 months of age, from 42 days to 90 days of age

Exclusion Criteria:

* Was born prior to 37 weeks of gestation.
* Has a history of invasive pneumococcal disease (IPD) (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV), any component of the licensed pediatric vaccines to be administered concomitantly in the study, or any diphtheria toxoid-containing vaccine.
* Has any contraindication to the concomitant study vaccines being administered in the study.
* Has external auditory canal atresia/stenosis.
* Has a known or suspected impairment of immunological function.

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7119 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a First Episode of Vaccine-Type Acute Otitis Media (VT-AOM) Caused by the Pneumococcal Serotypes Contained in V114 | Up to ~36 months
  The number of participants with VT-AOM will be presented.
Percentage of Participants with Serious Adverse Events | Up to ~36 months
  A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Percentage of Participants with Vaccine-Related Serious Adverse Events | Up to ~36 months
  A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Percentage of Participants Who Discontinued the Study due to Serious Adverse Events | Up to ~36 months
  A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Percentage of Participants Who Died | Up to ~36 months
  The percentage of participants who died from any cause during the study will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- Thailand (13):
  - Chulalongkorn University ( Site 0008), Bangkok, Bangkok
  - Phramongkutklao Hospital ( Site 0003), Bangkok, Bangkok
  - Siriraj Hospital ( Site 0004), Bangkok, Bangkok
  - Ramathibodi Hospital, Mahidol University ( Site 0009), Rajthevee, Bangkok
  - Bhumibol Adulyadej Hospital ( Site 0013), Sai Mai, Bangkok
  - Panyananthaphikkhu Chonprathan Medical Center ( Site 0014), Pak Kret, Changwat Nonthaburi
  - Faculty of Medicine Thammasat Univ. ( Site 0007), Khong Luang, Changwat Pathum Thani
  - Prince of Songkla University Faculty of Medicine ( Site 0005), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0001), Chiang Mai
  - Chiang Rai Prachanuchro Hospital-Pediatrics ( Site 0015), Chiang Rai
  - Srinagarind Hospital ( Site 0002), Khon Kaen
  - Bamrasnaradura Infectious Disease Institute ( Site 0011), Nonthaburi
  - Sappasit Prasong Hosptial-Pediatric ( Site 0016), Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com